CLINICAL TRIAL: NCT02518126
Title: Comparison of LIF (Leukemia Inhibitory Factor) Level Between Neonates Who Are IUGR (Intra Uterine Growth Restriction) and Those Who Are AGA (Average for Gestational Age)
Brief Title: Leukemia Inhibitory Factor Level in Intrauterine Growth Restriction Neonates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0176-15-RMB CTIL
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: to Compare LIF Level in Cord Blood of Embryo's That Are IUGR to Those That Are AGA
Keywords: LIF IUGR
MeSH Terms: interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood and a small peace of the placenta

GROUPS / COHORTS (2):
- control: Women with IUGR embryos so that their fetal weight estimate puts them in a percentile bellow 10th percentile
  Interventions: Other: blood sample and tissue sample
- IUGR: Women with AGA embryos so that their fetal weight estimate puts them in a percentile between 20th and 80th percentiles
  Interventions: Other: blood sample and tissue sample

INTERVENTIONS:
Other: blood sample and tissue sample — After birth and fetal umbilical cord disconnection, a blood sample will be taken from the umbilical cord (cord blood) of IUGR and of AGA fetuses (5cc) for cytokine ELISA testing. Also a small sample of the placenta will be examined in order to assess the level of ACTH protein in IUGR and AGA embryos

SUMMARY:
To see if there is a relationship between the level of LIF in IUGR fetuses and compared to the level of LIF in AGA fetuses

DETAILED DESCRIPTION:
During embryonic development, there are several cytokines such as: LIF (Leukemia inhibitory factor), ciliary neurotrophic factor (CNTF), epidermal growth factor family (EGF), neuregulin 1 (NRG1) and transforming growth factor β (TGFβ) that were found are associated with neurogenesis and differentiation of brain cells .

LIF is a cytokine that is essential for the development of the central nervous system, and has recently been shown in rats that maternal LIF stimulates placental ACTH that in turn promotes secretion of fetal LIF from nRBC , which in turn promotes brain development of the fetus Other studies on IUGR (Intra Uterine Growth Restriction) have shown that IUGR fetuses have more CP (Cerebral palsy) than those who were AGA (Average for Gestational Age) The hypothesis is that LIF is related to the proper development of the nervous system in the fetus and by testing cord blood of embryos IUGR and the placenta we will find changes in LIF and ACTH compared with AGA fetuses level.

Studies have also shown a relationship between CP and IUGR, but the mechanism for this relationship is unclear.

The purpose of our research is to see if there is a relationship between the level of LIF in IUGR fetuses and compared to the level of LIF in AGA fetuses, in one of two ways:

* Changes in the secretion of ACTH in placenta
* Changes in levels of LIF in the umbilical cord blood

ELIGIBILITY:
Inclusion Criteria:

* Women that the Fetal weight estimate puts the fetus bellow the 10th percentile and those that the fetal weight estimate are between 20th and 80th percentiles

Exclusion Criteria:

* Women who do not agree
* known Genetic diseases of abnormalities in the fetus

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women with fetuses who are AGA and those with fetuses that are IUGR
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
LIF Protein Level in IUGR Neonates vs. AGA neonates | 2 years